CLINICAL TRIAL: NCT02396927
Title: Three-dimensional High-definition (3DHD) Laparoscopy Versus Two-dimensional High-definition (2DHD) Laparoscopy in Cholecystectomy: a Clinical Controlled Randomized Double Blinded Trial.
Brief Title: 3D HD Versus 2D HD in Cholecystectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Herlev Hospital (Other)
Responsible Party: Principal Investigator, Charlotte Fergo, Miss, Herlev Hospital
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 3D_vs_2D_chol
Record Dates: First submitted 2015-03-12; First posted 2015-03-24 (Estimated); Last update posted 2017-02-28 (Actual); Status verified 2017-02

CONDITIONS: Cholelithiasis; Gall Bladder Disease
Keywords: 3D; Three-dimensional; laparoscopy; cholecystectomy
MeSH Terms: conditions — Cholelithiasis; Gallbladder Diseases

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 2D HD laparoscopy (Placebo Comparator): Elective laparoscopic cholecystectomy performed with the use of Olympus ENDOEYE FLEX in the 2DHD viewing mode
  Interventions: Device: 2D HD laparoscopy
- 3D HD laparoscopy (Active Comparator): Elective laparoscopic cholecystectomy performed with the use of Olympus ENDOEYE FLEX in the 3DHD viewing mode
  Interventions: Device: 3D HD laparoscopy

INTERVENTIONS:
Device: 3D HD laparoscopy — Olympus 3D laparoscopy ENDOEYE FLEX in high definition with the use of passive, polarizing glasses.
  Other Names: Olympus 3D ENDOEYE FLEX
  Arms: 3D HD laparoscopy
Device: 2D HD laparoscopy — Placebo
  Arms: 2D HD laparoscopy

SUMMARY:
The aim of this study is to compare 3D-laparoscopy versus 2D-laparoscopy with the use of HD resolution in cholecystectomy in terms of error rating, performance time and subjective assessment.

DETAILED DESCRIPTION:
Conventional laparoscopy can be very challenging, especially with the requirement of converting the two-dimensional image of the operating field to a three-dimensional perception. This can potentially lead to a detrimental effect on the learning curve as well for the feasibility of the operation for the more inexperienced surgeon. In our hospital, the high frequency of cholecystectomy serves as a basis for the minimally experienced surgeons to explore whether three-dimensional laparoscopy provides a better ability for solving complex intraoperative tasks than the conventional laparoscopy.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for elective cholecystectomy (out-patient treatment)

Exclusion Criteria:

* Previous upper abdominal surgery
* ASA-score 3 or above

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2015-03; Primary Completion 2017-09 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
Number of errors during the dissection of the Calot´s triangle | Expected duration: 20 minutes
  The unedited videos of the operations will be assessed according to GERT (Generic Error Rating Tool) by three surgeons, blinded to which optical modalities is used during the operations as done in a previous pilot study.

SECONDARY OUTCOMES:
Duration of the dissection of the Calot´s triangle | Expected duration: 20 minutes
Duration of surgery | Expected duration: 1 hour
The need for conversion to open surgery | intraoperative, expected duration of surgery: 1 hour
Estimated blood loss in ml | intraoperative, expected duration of surgery: 1 hour
Intraoperative complications | intraoperative, expected duration of surgery: 1 hour
  e.g. leakage of bile, leakage of gallstone, injury to the bile ducts, injury to organs.
Subjective assessment (Assessment of fatigue and perceived exertion) | an expected average of 15 minutes before and after the operation
  The surgeon will fill out questionnaires and scales.
Subjective assessment (optical modality and mental load assessment) | an expected average of 15 minutes after the operation
  The surgeon will fill out questionnaires and scales.

CONTACTS AND LOCATIONS:
Overall Officials: Charlotte Fergo, Principal Investigator — Herlev Hospital
Locations (1):
- Herlev Hospital, Herlev, Denmark

IPD SHARING:
Plan to Share IPD: No